CLINICAL TRIAL: NCT04265833
Title: Clinical, Radiographic and Histological Evaluation of Three Different Pulp Capping Materials in Indirect Pulp Treatment of Primary Teeth: A Randomized Clinical Trial
Brief Title: Evaluation of Three Different Pulp Capping Materials in Indirect Pulp Treatment of Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Merve AKCAY, assoc prof dr, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-1-TEZ-54
Record Dates: First submitted 2019-12-26; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Deep Caries
Keywords: deep caries; indirect pulp capping
MeSH Terms: interventions — tricalcium silicate; Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: randomized, three-arm parallel, two-blinded clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- calcium hydroxide (Active Comparator): Thirty six primary molar teeth with deep caries lesion were selected to apply indirect pulp therapy with calcium hydroxide. The carious peripheral dentin was removed at the enamel-dentin junction using a high-speed tungsten-carbide bur and the infected and necrotic soft dentin layer in the center was carefully removed to prevent pulp exposure. Cavity excavation was stopped when the residual dentin over the pulp tissue showed increased resistance to manual instrumentation, and the demineralized dentin (affected dentin) was left at the floor of the cavity.The residual demineralized dentin was covered with a thin layer of Ca(OH)2 (approximately 1 mm2) in accordance with the recommendations of the manufacturer. Afterwards capsule glass ionomer cement was placed on each capping material. Following the etching and bonding process, permanent restoration was finished with composite resin.
  Interventions: Other: Calcium hydroxide
- Biodentine (Experimental): Thirty seven primary molar teeth were selected to apply indirect pulp therapy with Biodentine. The carious peripheral dentin was removed at the enamel-dentin junction using a high-speed tungsten-carbide-bur and the infected and necrotic soft dentin layer in the center was carefully removed. Cavity excavation was stopped when the residual dentin over the pulp tissue showed increased resistance to manual instrumentation, and the demineralized dentin (affected dentin) was left at the floor of the cavity. A thin layer of tricalcium silicate-containing pulp-capping material (Biodentine) (approximately 1 mm2) consisting of powder and liquid was applied to the demineralized dentin tissue and a 12-min setting time was allowed for hardening, in accordance with the recommendations of the manufacturer. Afterwards capsule glass ionomer cement was placed on each capping material. Following the etching and bonding process, permanent restoration was finished with composite resin.
  Interventions: Other: Biodentine
- TheraCal LC (Experimental): Thirty six primary molar teeth with deep caries lesion were selected to apply indirect pulp therapy with TheraCal LC. The carious peripheral dentin was removed at the enamel-dentin junction using a high-speed tungsten-carbide bur and the infected and necrotic soft dentin layer in the center was carefully removed. Cavity excavation was stopped when the residual dentin over the pulp tissue showed increased resistance to manual instrumentation, and the demineralized dentin (affected dentin) was left at the floor of the cavity. Flowable form of resin-reinforced tricalcium silicate-containing material (TheraCal LC) was applied directly onto the demineralized dentin at a maximum thickness of 1 mm and was polymerized for 20 sec (Valo LED), in accordance with the recommendations of the manufacturer. Afterwards capsule glass ionomer cement was placed on each capping material. Following the etching and bonding process, permanent restoration was finished with composite resin.
  Interventions: Other: TheraCal LC

INTERVENTIONS:
Other: Biodentine — Biodentine has been shown to cause increased calcium ion release and this increase has been associated with the presence of pure tricalcium silicate and calcium chloride and the increased Ca(OH)2 formation
  Arms: Biodentine
Other: TheraCal LC — TheraCal LC (Bisco Inc, IL, USA) is a light-cured, resin-modified, calcium silicate-based material designed as a direct/indirect pulp-capping material. This agent has been shown to increase the pH on the pulpal surface thereby stimulating regenerative processes in the pulp, and ultimately contributing to the formation of dentin bridge
  Arms: TheraCal LC
Other: Calcium hydroxide — Calcium hydroxide (Ca[OH]2) is a successful pulp-capping agent activating the repair mechanism by stimulating the dentin-pulp complex. Ca(OH)2, with its bactericidal effects, protects the complex from bacterial effects and also has a stimulating effect on dentin remineralization
  Arms: calcium hydroxide

SUMMARY:
The aim of this randomized, controlled, three-arm parallel-group, double-blinded clinical trial was to evaluate the clinical, radiographic, and histopathological success of three different pulp-capping materials in one-stage indirect pulp treatment of primary teeth.

The study included a total of 109 patients aged 5-9 years who had primary teeth with deep carious lesions with or symptoms of irreversible pulpitis. The teeth were divided into three groups according to the pulp-capping agents: (I) Calcium hydroxide (Ca[OH]2) (control group) (n=36), (II) bioactive tricalcium silicate (Biodentine) (n=37), and (III) resin-based tricalcium silicate (TheraCal LC) (n=36). All the teeth were evaluated clinically and radiographically at postoperative months 6, 12, 18, and 24. A total of 23 primary mandibular second molars that were in their regular exfoliation period (24-40 months) were extracted and fixed in 10% formaldehyde solution. The specimens were evaluated histologically to assess the integrity of the odontoblastic layer, tertiary dentin formation and the quality of the dentin formed, severity of pulpitis, and other pulpal changes.

DETAILED DESCRIPTION:
Following the clinical and radiographic examinations, pulp vitality was assessed with cold thermal test (Chloraethyl; Wehr, Baden, Germany) and electrical pulp test. After local anesthesia injection, rubber-dam isolation was performed. In the first step of the IPC procedure, cavity preparation was performed and the caries were removed using a high-speed dental handpiece with a diamond bur. In the second step, the carious peripheral dentin was removed at the enamel-dentin junction using a high-speed tungsten-carbide bur and the infected and necrotic soft dentin layer in the center was carefully removed to prevent pulp exposure. Cavity excavation was stopped when the residual dentin over the pulp tissue showed increased resistance to manual instrumentation, and the demineralized dentin (affected dentin) was left at the floor of the cavity.

After this stage, the teeth were randomly divided into 3 groups:

Ca(OH)2 Group (Control): The residual demineralized dentin was covered with a thin layer of Ca(OH)2 (Dycal; Dentsply/Caulk, Dentsply International Inc. Milford, DE, USA) in accordance with the recommendations of the manufacturer.

Biodentine Group: A thin layer of tricalcium silicate-containing pulp-capping material (Biodentine, Septodont, France) consisting of powder and liquid was applied to the demineralized dentin tissue and a 12-min setting time was allowed for hardening, in accordance with the recommendations of the manufacturer.

TheraCal LC Group: Flowable form of resin-reinforced tricalcium silicate-containing material (TheraCal LC, Bisco Inc, IL, ABD) was applied directly onto the demineralized dentin at a maximum thickness of 1 mm and was polymerized for 20 sec (Valo LED, Ultradent Products Inc., South Jordan, USA), in accordance with the recommendations of the manufacturer.

Afterwards, in all three groups, capsule glass ionomer cement (Capsule; GC Corporation, Tokyo, Japan, Corporation, Tokyo, Japan) was placed on each capping material. Following the etching and bonding process, permanent restoration was finished with composite resin (Filtek Z250 Universal Restorative System, 3M ESPE Dental products, USA).

Histological examination A total of 23 primary mandibular second molars that were in their regular exfoliation period (in which the underlying permanent tooth germ had completed 2/3 of root formation) (24) and were found to be clinically and radiographically successful following IPC were extracted by the researcher and were processed for histological examination .All the extracted teeth were fixed in 10% formaldehyde solution. Three out of 23 specimens were excluded from the study since they were unsuitable for sectioning.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, vital and asymptomatic lower primary molars with deep caries lesions considered likely to result in pulp exposure if they were treated by a single and terminal excavation
* Positive pulp sensibility tested by an electric pulp tester and cold stimulation,
* Mild discomfort from chemical and thermal stimuli,
* Cooperative children and parents willing to follow the instructions and report for follow-up.

Exclusion Criteria:

* Signs of irreversible pulpitis (spontaneous pain, prolonged pain response etc.)
* The presence of percussion or palpation sensitivity, pathological mobility, or infection symptoms like fistula or abscess or discoloration in the clinical examination,
* Absence of normal lamina dura and periodontal range, presence of lesion, internal or external resorption or calcification in or around the root in the radiological examination,
* Children with special health care needs.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2015-02-08 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Clinical success rate of indirect pulp treatment | Change of clinical success from Baseline at 6 month
  Treatment is considered a clinical failure if one or more of the following signs are observed: Presence of tenderness to percussion or palpation, spontaneous pain or prolonged pain response, discoloration, infectious symptoms such as fistula or abscess, and pathological mobility. The treatment is regarded successful if clinical evaluation does not indicate any signs of failure.
Clinical success rate of indirect pulp treatment | Change of clinical success from baseline to 12 month
  Treatment is considered a clinical failure if one or more of the following signs are observed: Presence of tenderness to percussion or palpation, spontaneous pain or prolonged pain response, discoloration, infectious symptoms such as fistula or abscess, and pathological mobility. The treatment is regarded successful if clinical evaluation does not indicate any signs of failure.
Clinical success rate of indirect pulp treatment | Change of clinical success from baseline to 18 month
  Treatment is considered a clinical failure if one or more of the following signs are observed: Presence of tenderness to percussion or palpation, spontaneous pain or prolonged pain response, discoloration, infectious symptoms such as fistula or abscess, and pathological mobility. The treatment is regarded successful if clinical evaluation does not indicate any signs of failure.
Clinical success rate of indirect pulp treatment | Change of clinical success from baseline to 24 month
  Treatment is considered a clinical failure if one or more of the following signs are observed: Presence of tenderness to percussion or palpation, spontaneous pain or prolonged pain response, discoloration, infectious symptoms such as fistula or abscess, and pathological mobility. The treatment is regarded successful if clinical evaluation does not indicate any signs of failure.
Radiographic success rate of indirect pulp treatment | Change of radiographic success from baseline to 6 month
  For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The treatment is regarded successful if radiographic evaluation does not indicate any signs of failure.
Radiographic success rate of indirect pulp treatment | Change of radiographic success from baseline to 12 month
  For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The treatment is regarded successful if radiographic evaluation does not indicate any signs of failure.
Radiographic success rate of indirect pulp treatment | Change of radiographic success from baseline to 18 month
  For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The treatment is regarded successful if radiographic evaluation does not indicate any signs of failure.
Radiographic success rate of indirect pulp treatment | Change of radiographic success from baseline to 24 month
  For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The treatment is regarded successful if radiographic evaluation does not indicate any signs of failure.

SECONDARY OUTCOMES:
Histological success rate of indirect pulp treatment | up to 40 months (the teeth were extracted in regular exfoliation period (in which the underlying permanent tooth germ had completed 2/3 of root formation).
  For histologic evaluation, the treatment is rated as a failure when one or more of the following signs are present: absent of the integrity of the odontoblastic layer, absent of tertiary dentin formation, presence of pulpitis, presence of fibrosis and dystrophic calcification. The treatment is regarded successful if histologic evaluation does not indicate any signs of failure.

IPD SHARING:
Plan to Share IPD: No